CLINICAL TRIAL: NCT05452863
Title: Automatic Oxygen Supply With the O2matic Device for the Treatment of Hospitalized Heart Patients With Hypoxia
Brief Title: O2matic Cardiology Protocol
Acronym: O2matic-Card
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jens D Hove, MD,PHD, Associate Professor, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-19033702
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Diseases
Keywords: hypoxemia; cardiology; automatic oxygen supply
MeSH Terms: conditions — Heart Diseases; Hypoxia

STUDY DESIGN:
Intervention Model Description: Randomized, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic oxygen supply (Active Comparator): Oxygen will be supplied by the O2matic device
  Interventions: Device: O2matic administered oxygen
- Manual oxygen supply (Placebo Comparator): Oxygen will be supplied by nurse adjustments in the usual way
  Interventions: Device: Manual oxygen supply and adjustments

INTERVENTIONS:
Device: O2matic administered oxygen — Oxygen supply is adjusted from an almost continuous measurement of the oxygen saturation with an appropriate an previously tested algorithm.
  Arms: Automatic oxygen supply
Device: Manual oxygen supply and adjustments — Oxygen supply is adjusted from manual measurements of the oxygen saturation
  Arms: Manual oxygen supply

SUMMARY:
Automatic oxygen supply with the O2matic device has been shown to provided an enhanced oxygen treatment in patients with hypoxemia. O2matic was significantly better than manual control to maintain oxygen saturation within target interval and to reduce time with unintended hypoxemia in patients suffering from chronic obstructive pulmonary disease. This trial investigates the effect of using O2matic in hypoxic patients submitted to the Department of Cardiology.

DETAILED DESCRIPTION:
Oxygen supply to patients with cardiovascular disease has been subject to several investigations. Both too much and too little oxygen is supposed to be harmful. The O2matic device is a new way of supplying oxygen treatment which is significantly better than manual control to maintain oxygen saturation within target interval and to reduce time with unintended hypoxemia. The device has past favorable tests in patients suffering from chronic obstructive pulmonary disease. This study investigates the application of the O2matic device on hypoxic patients admitted to the Cardiology ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart disease and an oxygen saturation below 94% admitted to the Department of Cardiology
* Age of 30 or more
* Intellectual capacity to participate in the trial
* Willing to give informed accept of participation in the trial.

Exclusion Criteria:

* Unstable patients
* Need for ventilatory support except intermittent continuous positive airway pressure
* Fertile women (age<55 years) with a positive pregnancy test
* Unable to participate due to language or cognitive problems

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Time in designated saturation interval | 24 hours of treatment
  We have predefined an optimum saturation interval of 92-96% with a target of 93%

SECONDARY OUTCOMES:
Time with hypoxemia | 24 hours of treatment
  Time with saturation below 92% but above 85%
Time with severe hypoxemia | 24 hours of treatment
  Time with saturation below 85%
Time with hyperoxemia | 24 hours of treatment
  Time with saturation above 96%

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Hove, MD, PhD, Principal Investigator — Amager-Hvidovre Universitetshospital
Locations (1):
- Amager and Hvidovre Hospital University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen EF, Bech CS, Vestbo J, Andersen O, Kofod LM. Automatic oxygen titration with O2matic(R) to patients admitted with COVID-19 and hypoxemic respiratory failure. Eur Clin Respir J. 2020 Oct 14;7(1):1833695. doi: 10.1080/20018525.2020.1833695. PMID 33144929
- [Background] Kofod LM, Westerdahl E, Kristensen MT, Brocki BC, Ringbaek T, Hansen EF. Effect of Automated Oxygen Titration during Walking on Dyspnea and Endurance in Chronic Hypoxemic Patients with COPD: A Randomized Crossover Trial. J Clin Med. 2021 Oct 20;10(21):4820. doi: 10.3390/jcm10214820. PMID 34768338
- [Result] Hansen EF, Hove JD, Bech CS, Jensen JS, Kallemose T, Vestbo J. Automated oxygen control with O2matic(R) during admission with exacerbation of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 14;13:3997-4003. doi: 10.2147/COPD.S183762. eCollection 2018. PMID 30587955
- [Derived] Taraldsen IA, Grand J, Lukoschewitz JD, Seven E, Dixen U, Petersen M, Rytoft L, Jakobsen MM, Hansen EF, Hove JD. Automated oxygen administration versus manual control in acute cardiovascular care: a randomised controlled trial. Heart. 2024 Dec 13;111(1):27-34. doi: 10.1136/heartjnl-2024-324488. PMID 39486892
- [Derived] Taraldsen IA, Grand J, Lukoschewitz JD, Hansen EF, Hove JD. Automated versus manual oxygen administration for patients admitted with acute cardiovascular disease - a study protocol of a randomised controlled trial. Dan Med J. 2023 Mar 27;70(4):A12220784. PMID 36999819
- See also: Description of the device — https://o2matic.com